CLINICAL TRIAL: NCT06719453
Title: Prevalence of Alzheimer's Disease Pathology in a Large Norwegian Population-based Cohort and Predictive Power of Plasma p-tau217 and NfL.
Brief Title: Prevalence of Alzheimer's Disease Pathology in the Community
Acronym: HUNT4AD
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Göteborg University (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 3870
Record Dates: First submitted 2024-11-04; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-06

CONDITIONS: Dementia of Alzheimer Type; Alzheimer Disease; Mild Cognitive Impairment; Pathology; Biomarker in Early Diagnosis
Keywords: Blood-based markers; Population-based; p-tau217; cross-sectional; longitudinal; NfL; Alzheimer's disease pathology
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Trøndelag Health Study (The HUNT Study): (I) All participants from the HUNT4 70+ cohort (conducted 2017-2019, N=9,963) who have a blood sample (N=8,949). Participants underwent cognitive evaluation.
  (II) Selection of 3,948 participants from the HUNT3 cohort (conducted 2006-2008, n=8,548.). Selection criteria: Later participation in the HUNT4 70+ cohort or HUNT4 70+ AiT cohort and having an available blood sample in HUNT3. The 3,948 participants were further selected to include all those with a dementia diagnosis in HUNT4 70+ (N=approx. 1,100). Of the remaining HUNT3 participants included, 1/3 should have a diagnosis of normal cognition in HUNT4 70+, and 2/3 should have a diagnosis of mild cognitive impariment in HUNT4 70+.
  (III) All participants from the HUNT AiT cohort (Conducted 2021-2023, N=5,710) who have a blood sample. All HUNT4 70+ participants were invited to participate in HUNT4 AiT 4 years later. Participants underwent cognitive evaluation.

SUMMARY:
The goal of this observational study is to (I) study the proportion of people with Alzheimer's disease pathology in a large Norwegian population-based cohort of people aged 70 years or older and to (II) study longitudinal changes of Alzheimer's disease pathology in the same population over a 14 year period.

The main aims are:

* What is the proportion of people with Alzheimer's disease pathology, defined by elevated plasma p-tau217, in a large Norwegian population-based cohort of people aged 70 years or older.
* What is the proportion of people with Alzheimer's disease pathology, defined by elevated plasma p-tau217, among those with normal cognition, mild cognitive impairment and dementia in a large Norwegian population-based cohort of people aged 70 years or older.
* What is the association between plasma p-tau217 concentration and mild cognitive impairment or dementia 4, 10 and 14 years later, respectively.
* What is the association between plasma NfL concentration and mild cognitive impairment or dementia 4, 10 and 14 years later, respectively.

Data is used from The Nord-Trøndelag Health Study (HUNT) wave 3 (2006-2008) and 4 (2017 - 2019, also including HUNT AiT 2021-2023).

ELIGIBILITY:
Inclusion Criteria:

* Living in the area of Nord-Trøndelag, where the HUNT study is carried out.
* Age 70 or older when participating in HUNT4
* Available blood sample from HUNT3, HUNT4 70+ or HUNT4 70+ AiT

Exclusion Criteria:

* None

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The Nord-Trøndelag Health Study (HUNT) is carried out in the geographically defined area of Nord-Trøndelag i Norway and offers a good representation of the Norwegian population.
  The HUNT study has invited the adult population in the area to participate in four waves: HUNT1 (1984 - 1986), HUNT2 (1995-1997), HUNT3 (2006 - 2008) and HUNT4 (2017 - 2019). HUNT4 70+ also included a follow-up, Ageing in Trøndelag (AiT) (2021 - 2023). Notably, the HUNT4 study recruited all people 70 + years of age from HUNT4 to participate in the study, HUNT4 70+.
Sampling Method: Probability Sample
Enrollment: 9663 (Actual)
Dates: Start 2006-10-03 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Plasma p-tau217 and NfL concentrations in the HUNT4 70+ cohort, HUNT4 AiT cohort and in selected participants from HUNT3 | Biomarker concentration was measured in plasma samples from three time points: In the year 2006-2008, year 2017-2019 and year 2021-2023.
  Concentration of plasma p-tau217 measured by Alzpath217 and plasma NfL measured by Neurology 4-plex E kit. For p-tau217, we will administer a cut-off previously derived from the Wisconsin Registry for Alzheimer's Prevention study to define particpants as amyloid positive, amyloid negative or in an intermediate range.
Association between concentrations of plasma p-tau217 and NfL with cognitive status | Cognitive examination and blood sampling was conducted at two time points: In the year 2017-2019 and year 2021-2023.
  Association between concentrations of plasma p-tau217 and NfL with a clinical diagnosis of normal cognition, MCI and dementia in the HUNT4 70+ cohort and the HUNT4 AiT cohort
Predictive power of plasma p-tau217 and NfL | 14 years
  Reliability of plasma p-tau217 and NfL concentrations in HUNT3 and HUNT4 70+ for predicting cognitive impairment (I) measured by the MOCA in HUNT4 70+ and HUNT AiT, (II) defined by a clinical diagnosis of mild cognitive impairment or dementia in HUNT4 70+ and HUNT AiT.

SECONDARY OUTCOMES:
Association between kidney function and plasma p-tau217 | Cross-sectional measurements at three time points: In the year 2006-2008, year 2017-2019 and year 2021-2023. And longitudinal analysis (14 years, from 2006-2008 to 2021-2023))
  What is the association between eGFR and plasma p-tau217 concentration in a large population-based cohort of older adults.
Prevalence of amyloid pathology in different ApoE ε genotype groups | Plasma p-tau217 was measured in plasma samples at three time points: In the year 2006-2008, year 2017-2019 and year 2021-2023.
  Proportion of study participants in HUNT4 70+ and HUNT4 AiT with amyloid pathology according to plasma p-tau217 in different ApoE ε genotype groups.
  Proportion of participants with amyloid pathology according to plasma p-tau217 among selected study participants in HUNT3 aged 60 to 69 years at study participation, differentiated by ApoE ε genotype groups.
  ApoE ε genotype status in participants has already been previously established.

IPD SHARING:
Plan to Share IPD: Undecided
All researchers can apply for data at the HUNT research data senter.